CLINICAL TRIAL: NCT04954612
Title: Musculoskeletal Problems and Associated Factors in Children Aged Between 6-13 Years During the COVID-19 Pandemic
Brief Title: Musculoskeletal Problems in School Children During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/205
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Children; Musculoskeletal Disorder
Keywords: COVID-19; Remote education; Ergonomics
MeSH Terms: conditions — Musculoskeletal Diseases; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire study (Cross-sectional analytical clinical research) — Questionnaire study (Cross-sectional analytical clinical research)

SUMMARY:
During COVID-19 pandemic, in the lockdown period, reduced physical activity and obesity were reported in children.

In Turkey, face to face education was ceased after March 16, till the end of the previous academic year and education was tried to be substituted remotely.

A temporary lockdown was implemented for children and young people under the age of 20, between April 3 and June 5 2020. At 45 days following the lockdown of children, 72% of the parents with children aged 6-13 years stated that their screen time had increased to a mean of 6.4 hours per day.

Engaging more time in physical activity, and less in sedentary and leisure screen time was found to be associated with less anxiety during pandemic.

Before 2020-2021 academic year, government and educators increased their preparedness for the second and third waves and improved the technological infrastructure. Depending on grades, preferences of the family, primary education continued remotely between November 2020 and July 2021.

The aim of this study is to investigate whether musculoskeletal complaints are increased in school-age children during the pandemics and whether there is a relationship between the decreased level of physical activity, increased screen time, poor posture and musculoskeletal complaints.

DETAILED DESCRIPTION:
A survey assessing musculoskeletal pain in children in the last 1 month, and associated factors including presence of non-ergonomic postures during online education was structured by two physiatrists and a public health specialist after the review of the relevant literature. Several paediatric pain and musculoskeletal assessment tools were reviewed.

The survey consisted of a total of 66 questions including sociodemographic characteristics of the children and family (17 items), education hours, used technological device (7 items), screen time and physical activity (5 items), presence of musculoskeletal pain (27 items) and ergonomics (10 items).

Questions regarding the musculoskeletal pain were constructed based on The Nordic musculoskeletal questionnaire extended version (NMQ-E) which was translated and validated into Turkish. Pain or discomfort questions experienced in the nine body parts with binary choices (yes or no) were used. The figure in NMQ-E was used to describe body regions (the neck, shoulder, upper back, elbow, wrist/hand, low back, hip/ thigh, knee, ankle/foot) and pain questions were structured accordingly on this body diagram.

The questionnaire was created using the Qualtrics program. The survey was piloted among ten participants to ensure its readability and ease of completion. After obtaining permissions from Ministry of National Education of Turkey, survey link was shared with the school principles so that they distributed the survey to the guardians of children via smart phones or email. The survey will be available during two months and a reminder will be sent once a week.

ELIGIBILITY:
Inclusion Criteria:

* Being parent or guardian of a child between the ages of 6-13 years
* Having access to the Internet
* Being literate
* Giving consent to participate in the study

Exclusion Criteria:

* Children going to special education school

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A sample size of 1225 participants was calculated by assuming a musculoskeletal pain prevalence of 15% among children between the ages 6-13, with a confidence limit of 95% with a margin of error 2%.
Sampling Method: Probability Sample
Enrollment: 1225 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-09 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of musculoskeletal pain | One day
  Presence of musculoskeletal pain in one of the nine body parts

CONTACTS AND LOCATIONS:
Overall Officials: Özden Özyemişçi Taşkıran, Prof, Principal Investigator — Koc University School of Medicine Department of Physical Medicine and Rehabilitation; Sibel Sakarya, Prof, Study Director — Koc University School of Medicine Department of Infectious Disease; Zeynep Turan, Study Chair — Koc University School of Medicine Department of Physical Medicine and Rehabilitation; Esra Giray, Assoc Prof, Study Chair — Koc University School of Medicine Department of Physical Medicine and Rehabilitation
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Result] Kamper SJ, Henschke N, Hestbaek L, Dunn KM, Williams CM. Musculoskeletal pain in children and adolescents. Braz J Phys Ther. 2016 Feb 16;20(3):275-84. doi: 10.1590/bjpt-rbf.2014.0149. PMID 27437719
- [Result] Alaca N, Safran EE, Karamanlargil AI, Timucin E. Translation and cross-cultural adaptation of the extended version of the Nordic musculoskeletal questionnaire into Turkish. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):472-481. PMID 31789298
- [Result] Simons LE, Smith A, Ibagon C, Coakley R, Logan DE, Schechter N, Borsook D, Hill JC. Pediatric Pain Screening Tool: rapid identification of risk in youth with pain complaints. Pain. 2015 Aug;156(8):1511-1518. doi: 10.1097/j.pain.0000000000000199. PMID 25906349
- [Result] Gariepy G, McKinnon B, Sentenac M, Elgar FJJCIR. Validity and reliability of a brief symptom checklist to measure psychological health in school-aged children. 2016;9(2):471-484.
- [Result] Lauridsen HH, Hestbaek L. Development of the young spine questionnaire. BMC Musculoskelet Disord. 2013 Jun 12;14:185. doi: 10.1186/1471-2474-14-185. PMID 23758965
- [Result] Majumdar P, Biswas A, Sahu S. COVID-19 pandemic and lockdown: cause of sleep disruption, depression, somatic pain, and increased screen exposure of office workers and students of India. Chronobiol Int. 2020 Aug;37(8):1191-1200. doi: 10.1080/07420528.2020.1786107. Epub 2020 Jul 13. PMID 32660352
- [Result] Robbins M, Johnson I, Cunliffe CJCC. Encouraging good posture in school children using computers. 2009;12(1):35-44.
- [Result] Tan A, Strauss VY, Protheroe J, Dunn KM. Epidemiology of paediatric presentations with musculoskeletal problems in primary care. BMC Musculoskelet Disord. 2018 Feb 6;19(1):40. doi: 10.1186/s12891-018-1952-7. PMID 29409492